CLINICAL TRIAL: NCT00236132
Title: " A Multicenter Study Comparing the Clinical Outcomes of the Nuss and Ravitch Procedures for Repair of Pediatric Pectus Excavatum"
Brief Title: "A Multicenter Study Comparing the Clinical Outcomes of the Nuss and Ravitch Procedures for Repair Of Pediatric Pectus Excavatum
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Children's Health System, Inc. (Other)
Collaborators: Walter Lorenz Surgical Corporation (Unknown)
Other Study IDs: IRB #01-02-FB-0032; NCT00275470 (obsolete NCT alias)
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Last update posted 2007-10-12 (Estimated); Status verified 2007-10

CONDITIONS: Repair of Pectus Excavatum

SUMMARY:
The main goal of the pectus multicenter outcomes study is to document the utility of PEx repair in improving health and quality of life and to test the prevailing belief that the two predominant surgical procedures currently in use for PEx repair are essentially equivalent in terms of long-term outcomes.

We believe the uncertainty about the impact of PEx on cardiopulmonary function is due to part to the fact that the previous studies have not measured the physiological parameters mostly likely affected by the defect. A protocol to test this was developed. Thus, we propose to use these measures as well as conventional output of progressive exercise test to examine cardiopulmonary function before and after surgical repair of PEx within the context of the original study.

ELIGIBILITY:
Inclusion Criteria:Haller index by thoracic computed tomography (CT) scan of 3.2 or greater, has decided to have surgery to repair PEx, Written informed consent obtained from the parent or guardian of the subject,or, fro subjects 18-21 years, from the subject him(her)self, and assent of the child.

-

Exclusion Criteria:Pectus carinatum, Poland's syndrome or other comlex chest wall anomaly,Previous repair of PEx by any technique, Previous thoracic surgery, Congenital heart disease, Bleeding dyscrasia, History of major anesthetic risk factors such as malignant hyperthermia, Pregnancy, Surgical repair to be performed with bar other than stainless steel.

-

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 360 (Estimated)
Dates: Start 2001-08; Study Completion 2008-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Kelly, Jr., MD, Principal Investigator — Children's Hospital of The King's Daughters
Locations (12):
- United States (11):
  - Yale New Haven Children's Hospital, New Haven, Connecticut
  - All Children's Hospital, St. Petersburg, Florida
  - Kapi'olani Medical Center for Women and Children, Honolulu, Hawaii
  - John Hopkins Hospital, Baltimore, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Children's Hospital of New York -Presbyterian, New York, New York
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Medical Center Dallas, Dallas, Texas
  - Childern's Hospital of The King's Daughters, Norfolk, Virginia
  - Children's Hospital Of Wisconsin, Milwaukee, Wisconsin
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Kelly RE Jr, Mellins RB, Shamberger RC, Mitchell KK, Lawson ML, Oldham KT, Azizkhan RG, Hebra AV, Nuss D, Goretsky MJ, Sharp RJ, Holcomb GW 3rd, Shim WK, Megison SM, Moss RL, Fecteau AH, Colombani PM, Cooper D, Bagley T, Quinn A, Moskowitz AB, Paulson JF. Multicenter study of pectus excavatum, final report: complications, static/exercise pulmonary function, and anatomic outcomes. J Am Coll Surg. 2013 Dec;217(6):1080-9. doi: 10.1016/j.jamcollsurg.2013.06.019. PMID 24246622
- [Derived] Kelly RE Jr, Cash TF, Shamberger RC, Mitchell KK, Mellins RB, Lawson ML, Oldham K, Azizkhan RG, Hebra AV, Nuss D, Goretsky MJ, Sharp RJ, Holcomb GW 3rd, Shim WK, Megison SM, Moss RL, Fecteau AH, Colombani PM, Bagley T, Quinn A, Moskowitz AB. Surgical repair of pectus excavatum markedly improves body image and perceived ability for physical activity: multicenter study. Pediatrics. 2008 Dec;122(6):1218-22. doi: 10.1542/peds.2007-2723. PMID 19047237